CLINICAL TRIAL: NCT01339585
Title: The Effect of Timing of Transcranial Direct Current Stimulation (tDCS) for Enhancing Learning During Cognitive Training
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The University of New South Wales (Other)
Responsible Party: Principal Investigator, Melissa Pigot, Research Assistant, The University of New South Wales
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Basic Science
Other Study IDs: HREC 11064
Record Dates: First submitted 2011-04-01; First posted 2011-04-20 (Estimated); Last update posted 2014-08-12 (Estimated); Status verified 2014-08

CONDITIONS: Effects on Learning
MeSH Terms: interventions — Transcranial Direct Current Stimulation

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Timing of tDCS (Experimental)
  Interventions: Device: Transcranial direct current stimulation (tDCS)
- Alternative timing of tDCS (Experimental)
  Interventions: Device: Transcranial direct current stimulation (tDCS)

INTERVENTIONS:
Device: Transcranial direct current stimulation (tDCS) — Eldith Direct Current Stimulator (NeuroConn GmbH, Germany)

SUMMARY:
This project will investigate a novel strategy for enhancing cognitive training (CT). Specifically, the investigators aim to combine a non-invasive form of brain stimulation (tDCS) with CT. This study will examine the optimal time interval - whether tDCS should be administered either before or during CT.

ELIGIBILITY:
Inclusion Criteria:

* Participants will be healthy right-handed subjects aged 18 to 40 years.

Exclusion Criteria:

* Concurrent medication likely to affect mental performance,
* Current history of drug or alcohol abuse or dependence,
* Any psychiatric or neurological disorder,
* Recent head injury, or history of seizure or stroke.

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2011-05; Primary Completion 2014-05 (Actual)

PRIMARY OUTCOMES:
Change in performance across each condition. | Over 2 days, with each condition conducted 1 month apart.
  D prime, number of correct responses, and number of errors.

CONTACTS AND LOCATIONS:
Locations (1):
- School of Psychiatry, Sydney, New South Wales, Australia